CLINICAL TRIAL: NCT04118829
Title: Correlation of Serum Level of Perampanel (PER) Level to Cerebrospinal Fluid (CSF) Levels of PER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Aashit Shah, Chief of Neurology, Carilion Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-19-347
Record Dates: First submitted 2019-09-16; First posted 2019-10-08 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Epilepsy; Seizures
Keywords: Perampanel
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group one (Experimental): The Group 1 patients will be taking PER up to 14 days following surgical intervention as per discretion of the treating neurosurgeon.
  Interventions: Drug: Perampanel
- Group Two (Experimental): The Group 2 patients will be taking PER as part of their maintenance AED regimen and will continue on the same maintenance dosage postoperatively.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — For group 1 the PER dose will be administered 2-14 hours prior to sample collection. They will be administered a single dose of PER (8 mg, 12 mg or 16 mg) followed by 4 mg/day for 14 days starting on postoperative day 1 (if continued prophylaxis with PER is needed).
  It is anticipated that patients in group 2 will have the daily dose of PER in these individuals will range from 4 - 12 mg/day.

SUMMARY:
Perampanel is a drug used to treat patients with epilepsy/seizures. This study is designed to determine how much perampanel actually crosses the blood brain barrier into the cerebral spinal fluid when the drug is taken.

DETAILED DESCRIPTION:
Perampanel is a drug used to treat patients with epilepsy/seizures. This study is designed to determine how much perampanel actually crosses the blood brain barrier into the cerebral spinal fluid when the drug is taken.

During a routinely scheduled neurosurgical procedure, one to two mL of cerebral spinal fluid will be obtained from the subarachnoid space of the brain. Five mL of arterial blood will also be drawn from the patients arterial line during their procedure. The blood samples and cerebral spinal fluid samples will be compared to see how much perampanel is in the blood versus the cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years-old) who are scheduled to undergo brain surgery and need antiepileptic medication for prophylaxis or treatment of seizures
* Able to provide informed consent

Exclusion Criteria:

* Patient unable to provide informed consent
* Allergy to PER or its component
* Patient with significant renal (creatinine clearance 35 ml/min) or hepatic impairment
* Pregnant or lactating females will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Blood brain barrier serum levels | 3 weeks
  To determine the blood brain barrier(BBB) penetration of PER by measuring ratio of serum level to that of CSF measured on simultaneously obtained samples

CONTACTS AND LOCATIONS:
Overall Officials: Aashit Shah, MD, Principal Investigator — Physician
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
We will not share any individual participant data. Data analysis will involve aggregated data.